CLINICAL TRIAL: NCT06933680
Title: The Effect of Sphenopalatine Ganglion Block on Intraoperative Analgesia, Postoperative Edema, and Pain in Bimaxillary Orthognathic Surgery
Brief Title: Sphenopalatine Ganglion Block in Bimaxillary Orthognathic Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Büşra Ceylan, Resident Physician in Anesthesiology and Reanimation, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: BezmialemVU-AR-BC-01
Record Dates: First submitted 2025-03-27; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Bimaxillar Surgery; Sphenopalatine Ganglion Block
Keywords: sphenopalatine ganglion block; pain; bimaxillary orthognathic surgery; edema; swelling
MeSH Terms: conditions — Pain; Edema | interventions — Sphenopalatine Ganglion Block

STUDY DESIGN:
Intervention Model Description: For the study's randomization, 50 sealed envelopes were prepared. Inside, 25 envelopes were labeled "SPG group" and 25 were labeled "control group." One sealed envelope is randomly selected and given to the anesthesia technician.
  The anesthesia technician prepares either Marcaine or saline solution for the block and hands it to the anesthesiologist without revealing its contents. The anesthesia technician also assigns a number to each patient based on their registration order and records the patient's group in a confidential list.
  The anesthesiologist, who is blinded to the group assignments, performs the block and monitors the patient, records. The surgical team, also blinded, evaluates surgical comfort. Patients remain blinded to their group during follow-ups.
  At the end of the study, patient data will be matched with their assigned groups for analysis.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPG block group (Active Comparator): This group will receive a SPG block using 4 ml of 5% bupivacaine after entübastion.
  Interventions: Procedure: Sphenopalatine Ganglion Block
- control group (Sham Comparator): This group will receive a sham block using the same method using 4 ml of physiological saline after intubation.
  Interventions: Procedure: Sham Block

INTERVENTIONS:
Procedure: Sphenopalatine Ganglion Block — To perform an SPG block, the ultrasound linear probe is placed parallel to the zygomatic bone, facing anteriorly, to obtain an image that includes the ramus of the maxilla and mandible and the pterygoid process of the sphenoid bone.
  A 23-gauge, 50 mm needle is inserted just behind the posterior orbital rim and advanced in an antero-caudal direction over the zygomatic arch. When the needle reaches the pterygopalatine fossa at approximately 5 cm, aspiration is performed to check for blood. If no blood is seen, 4 mL of 0.5% bupivacaine is injected.
  The procedure is performed on both sides
  Other Names: Meckel ganglion block; pterygopalatine ganglion block
  Arms: SPG block group
Procedure: Sham Block — To perform a Sham block, the ultrasound linear probe is placed parallel to the zygomatic bone, facing anteriorly, to obtain an image that includes the ramus of the maxilla and mandible and the pterygoid process of the sphenoid bone.
  A 23-gauge, 50 mm needle is inserted just behind the posterior orbital rim and advanced in an antero-caudal direction over the zygomatic arch. When the needle reaches the pterygopalatine fossa at approximately 5 cm, aspiration is performed to check for blood. If no blood is seen, 4 mL of %0,9 NaCl is injected.
  The procedure is performed on both sides.
  Arms: control group

SUMMARY:
The goal of this clinical trial is to evaluate whether sphenopalatine ganglion (SPG) block helps with intraoperative pain control, reduces postoperative edema, and decreases pain in adults aged 18 to 45 undergoing bimaxillary orthognathic surgery.

The main questions it aims to answer are:

* Does SPG block help decrease postoperative swelling and pain compared to a sham block?
* Does it improve pain control during surgery and reduce opioid use? Researchers will compare patients receiving SPG block to those receiving a sham block to determine if this technique provides better pain relief and reduces postoperative complications.

Participants will:

* Be 18 to 45 years old and undergo bimaxillary orthognathic surgery.
* Be randomly assigned to receive either a SPG block or a sham block before surgery.
* Be monitored for 1 month after surgery to assess pain levels, swelling, opioid use, and possible complications.

DETAILED DESCRIPTION:
Orthognathic surgery is a procedure used to correct jaw bone problems that are present from birth or develop over time. During this surgery, multiple cuts, tissue separation, and bone reshaping (osteotomy) are done on the upper and lower jaw. After the surgery, the body responds with an inflammatory reaction, causing edema and pain. As the tissues heal, the edema and pain gradually decrease.

Edema is a common result of orthognathic surgery and can affect recovery time, return to normal activities, and hospital stay. Research shows that reducing edema can improve a patient's quality of life. Excessive edema can also cause pain and discomfort. To manage this, treatments such as steroids, laser therapy, lymphatic drainage massage, and cold applications are used.

The SPG is a nerve center that contains both sensory and autonomic nerve fibers. It connects to the trigeminal nerve, facial nerve, internal carotid plexus, and superior cervical ganglion. The SPG plays a role in widening brain blood vessels, providing sensation to the soft palate, tonsils, upper lip, and mouth floor, and controlling tear gland secretions.

In our study, it is anticipated that SPG block may help prevent intraoperative abnormal hemodynamic changes (by facilitating the control of heart rate and mean arterial pressure), reduce bleeding, decrease anesthetic drug consumption, lower the incidence of postoperative nausea and vomiting, and improve postoperative pain control and edema reduction. As a result, the postoperative comfort of patients undergoing orthognathic surgery can be enhanced with a cost-effective and easily applicable method, potentially reducing the risk of chronic pain in the long term. Additionally, by minimizing surgery-related edema and jaw muscle spasms, patients may achieve an optimal quality of life more quickly. Due to the limited number of studies on this technique in oral and maxillofacial surgery, our study is expected to pave the way for future research in this area.

ELIGIBILITY:
Inclusion Criteria:

* Patients with bimaxillary orthognathic surgery indication
* Patients with American Society of Anesthesiologistsscores (ASA) I-II
* Patients between the ages of 18-45

Exclusion Criteria:

* Patients with local anesthetic allergy
* Patients undergoing genioplasty
* Syndromes associated with secondary deformities in addition to jaw deformities
* Patients with a history of jaw surgery
* Patients with uncontrolled hypertension
* Patients with a history of substance abuse
* Patients with chronic pain lasting more than 3 months
* Patients using analgesic and hypnotic agents for more than 2 weeks
* Recent situations that may cause facial edema (tooth extraction, facial trauma, etc.)
* Patients with psychiatric disorders
* Patients with diabetes mellitus
* Patients with bleeding disorders

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Postoperative Edema | Measurements are taken preoperatively, at 24 hours postoperatively, on postoperative day 3, day 7 and at 1 month.
  Using the technique of Gabka and Matsumura, gonion, mentum, and tragus are marked with methylene blue before surgery. The distances between the marks are measured bilaterally in millimeters using a flexible ruler and recorded.
  The measurement points will include:
  * Tragus-labial commissure distance
  * Tragus-alar notch distance
  * Gonion-lateral canthus distance
  * Tragus-mentum distance
  Postoperatively, edema measurements are taken from the same points.
Postoperative Pain | The patient's pain at rest and during movement is evaluated at 30 minutes, 6 hours, 12 hours, 24 hours and 48 hours following the end of the surgery.
  The numeric rating scale(NRS) is used to evaluate postoperative pain. Patients are asked to rate their pain on the scale of 0 to 10, with 0 indicating no pain and 10 indicating unbearable pain. Nrs scores are recorded.

SECONDARY OUTCOMES:
Effect of the Block on Temperature | Measurements are taken every 5 minutes for the first 1 hour after induction.
  Starting before the block, the forehead skin temperature will be recorded every 5 minutes for 1 hour. During this period, the block time and surgical draping time are noted.
Heart rate | Measurements are taken every 15 minutes preoperatively and throughout the surgery
  Heart rate is monitored and recorded perioperatively using noninvasive monitoring.
Mean arterial pressure | Measurements are taken every 15 minutes preoperatively and throughout the surgery
  Mean arterial pressure is monitored and recorded perioperatively using noninvasive monitoring.
Opioid and Anesthetic Agent Consumption | The agents used during surgery are recorded once at the end of anesthesia.
  The amount of sevoflurane required to maintain the bispectral index (BIS) value within the target range and the total remifentanil used are recorded at the end of each patient's surgery.
Quality of the surgical field | That is recorded once at the end of surgery.
  The surgeon assesses the quality of the surgical field using a predefined category scale, adapted from Fromme GA et al. at the end of the surgery.
  Fromme Scale :
  * Grade 1: Massive uncontrollable bleeding
  * Grade 2: Bleeding, heavy but controllable, that significantly interferes with dissection
  * Grade 3: Moderate bleeding that moderately compromises surgical dissection
  * Grade 4: Moderate bleeding, a nuisance but without interfering with aaccurate dissection
  * Grade 5: Bleeding, so mild it was not even a surgical nuisance
  * Grade 6: No bleeding, virtually bloodless field
Postoperative Analgesic Consumption | These assessments are recorded at 30 minutes, 6 hours, postoperative day 1, day 2 and day 3.
  As a secondary parameter for pain assessment, the amount of opioid analgesic (tramadol) used, the number of requests and the need for rescue analgesics are recorded through patient-controlled analgesia devices.
Mouth Opening | Measurements are taken preoperatively, on postoperative day 1, day 3, and day 7.
  The distance between font teeth is measured and recorded with soft ruler.
Nausea and Vomiting | These assessments are recorded at 30 minutes, 6 hours, postoperative day 1, day 2 and day 3.
  Nausea and vomiting are evaluated using a 4-point categorical scale 0 = No nausea
  1. = Nausea only
  2. = Nausea with retching
  3. = Vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Büşra Ceylan, Resident Doctor, Principal Investigator — Bezmialem Vakıf Üniversitesi; Harun Uysal, Associate Professor, Study Director — Bezmialem Vakıf Üniversitesi; Ayda Türköz, Professor Doctor, Study Director — Medipol Acıbadem District Hospital
Locations (1):
- Bezmialem Vakıf Üniversitesi, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith CR, Dickinson KJ, Carrazana G, Beyer A, Spana JC, Teixeira FJP, Zamajtuk K, Maciel CB, Busl KM. Ultrasound-Guided Suprazygomatic Nerve Blocks to the Pterygopalatine Fossa: A Safe Procedure. Pain Med. 2022 Aug 1;23(8):1366-1375. doi: 10.1093/pm/pnac007. PMID 35043949
- [Background] Sumphaongern T, Chantarangsu S. Effect of Dexmedetomidine on Blood Loss and Patient Outcomes in Orthognathic Surgery: A Randomised Clinical Trial. Int Dent J. 2025 Jun;75(3):1961-1969. doi: 10.1016/j.identj.2025.01.009. Epub 2025 Jan 28. PMID 39880716
- [Background] Keyhan SO, Fallahi HR, Cheshmi B, Mokhtari S, Zandian D, Yousefi P. Use of piezoelectric surgery and Er:YAG laser:which one is more effective during impacted third molar surgery? Maxillofac Plast Reconstr Surg. 2019 Aug 6;41(1):29. doi: 10.1186/s40902-019-0212-6. eCollection 2019 Dec. PMID 31448247
- [Background] Sari N, Uysal E. Endoscopic Sphenopalatine Ganglion Block Efficacy in the Management of Periorbital Edema and Ecchymosis After Septorhinoplasty. J Craniofac Surg. 2021 May 1;32(3):983-987. doi: 10.1097/SCS.0000000000007189. PMID 33055565
- [Background] Robiony M, Demitri V, Costa F, Politi M, Cugini U. Truncal anaesthesia of the maxillary nerve for outpatient surgically assisted rapid maxillary expansion. Br J Oral Maxillofac Surg. 1998 Oct;36(5):389-91. doi: 10.1016/s0266-4356(98)90653-2. PMID 9831062
- [Background] Shah RJ, Dixon B, Padalia D. Sphenopalatine Ganglion Radiofrequency Thermocoagulation. 2023 Jul 7. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK536944/ PMID 30725629
- [Background] Dominguez Camacho A, Velasquez SA, Benjumea Marulanda NJ, Moreno M. Photobiomodulation as oedema adjuvant in post-orthognathic surgery patients: A randomized clinical trial. Int Orthod. 2020 Mar;18(1):69-78. doi: 10.1016/j.ortho.2019.09.004. Epub 2019 Oct 31. PMID 31678060